CLINICAL TRIAL: NCT06405893
Title: What Makes People Better at Naming Pictured Objects
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Lori James, Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-049
Record Dates: First submitted 2024-05-04; First posted 2024-05-09 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Healthy Aging
Keywords: Aging; Mindfulness; Speech Production

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Breathing (Experimental): 10 minute mindful breathing exercise
  Interventions: Behavioral: Mindful breathing exercise
- Control (Sham Comparator): 10 minute recorded info about mindfulness
  Interventions: Behavioral: Mindful breathing exercise

INTERVENTIONS:
Behavioral: Mindful breathing exercise — Participants do a 10 minute guided mindful breathing exercise or participants do listen to a 10 minute control recording

SUMMARY:
This study is being conducted to learn more about how mindful breathing might be related to the ability to produce names for pictured objects. Participants will engage with an exercise about mindful breathing or an auditory presentation and then name pictured objects as quickly as they can. They will also complete some surveys and other measures and wearing equipment on their finger to monitor their heart rate throughout the study. Participation will take approximately 1 hour.

DETAILED DESCRIPTION:
This study is being conducted to learn more about how mindful breathing might be related to the ability to produce names for pictured objects. Up to 200 participants between ages 18-35 or 60-80 who are native, fluent speakers of English will engage with an exercise about mindful breathing or an auditory presentation. They will then name pictured objects as quickly as they can. Sessions will be audio recorded for later scoring. Participants will also complete demographics forms, a vocabulary test, and a measure of their current anxiety. Those over age 60 will also complete a cognitive function assessment. Participants will be wearing equipment on their finger to monitor their heart rate throughout the study. Participation will take approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-35 or 60-80
* Fluent English speaker

Exclusion Criteria:

* Younger than 18 years old
* Between ages 36-59
* Older than age 80
* Not a fluent English speaker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Response Accuracy for Naming Pictures (% correct) | Under 1 hour
  Percent of valid trials on which correct object names were provided will be computed. The measure was designed for use in this study.
Response Time for Naming Pictures (onset time in ms) | Under 1 hour
  Mean response onset time for valid trials on which correct object names were provided will be computed. The measure was designed for use in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- UCCS, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual data as of now. If the study is submitted for publication to a journal that requires it, data will be made available.